CLINICAL TRIAL: NCT00399581
Title: Phase II Clinical Trial of Two Approaches to High Frequency Oscillatory Ventilation in Acute Respiratory Distress Syndrome
Brief Title: Comparison of Two Methods of High Frequency Oscillatory Ventilation in Individuals With Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Roy Brower, MD, Professor of Medicine, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 471; P50HL073994 (NIH)
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2009-07

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; Mechanical Ventilation; Lung
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFOV-Lo (Experimental): High Frequency Oscillatory Ventilation using lower mean airway pressures and higher FiO2s.
  Interventions: Procedure: High Frequency Oscillatory Ventilation-Lo
- HFOV-Hi (Experimental): High Frequency Oscillatory Ventilation using higher mean airway pressures
  Interventions: Procedure: High Frequency Oscillatory Ventilation-Hi

INTERVENTIONS:
Procedure: High Frequency Oscillatory Ventilation-Hi — HFOV will be conducted with recruitment maneuvers and with a table of mPaw and FiO2s that include higher mPaw's.
  Arms: HFOV-Hi
Procedure: High Frequency Oscillatory Ventilation-Lo — HFOV will be conducted without routine recruitment maneuvers and with a table of mPaw and FiO2s that include relatively low mPaw's.
  Arms: HFOV-Lo

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe lung condition that causes respiratory failure. Individuals with ARDS often require the use of an artificial breathing machine, known as a mechanical ventilator. High frequency oscillatory ventilation (HFOV) is a form of mechanical ventilation that pumps small amounts of air into the lungs at a constant high rate. The purpose of this study is to compare the safety and efficacy of two HFOV methods in individuals with ARDS.

DETAILED DESCRIPTION:
ARDS is a serious condition that involves lung inflammation and fluid accumulation in the air sacs, leading to low blood oxygen levels and respiratory failure. It is often fatal and affects approximately 160,000 individuals each year in the United States. The main form of treatment for ARDS is delivery of oxygen and a continuous level of pressure to the damaged lungs through mechanical ventilation. However, some methods of mechanical ventilation may cause ventilator-associated lung injury (VALI), a condition that can result from overdistension of the lungs during inspiration or from excessive mechanical forces. VALI can delay or prevent healing from respiratory failure.

HFOV is a mechanical ventilation method that pumps small amounts of air into the lungs at a constant high rate. Because the increments of air are small the likelihood of experiencing overdistension and developing VALI may be reduced. While HFOV is an effective, commonly used ventilation method, there have been no studies that demonstrate the efficacy of HFOV in comparison to the efficacy of conventional mechanical ventilation methods. This study will compare two different HFOV techniques: the HFOV-Hi method, which uses higher airway pressure, and the HFOV-Lo method, which uses lower airway pressure. The purpose of this study is to compare the safety and efficacy of HFOV-Hi, HFOV-Lo, and standard mechanical ventilation methods in individuals with ARDS.

This study will enroll individuals with ARDS at four Baltimore hospitals. Participants will be randomly assigned to receive either HFOV-Hi or HFOV-Lo. All participants will receive their assigned HFOV method for 7 days, until spontaneous breathing occurs, or until death, whichever occurs first. Blood collected at baseline and Days 1 and 3 will be analyzed for markers of inflammation and lung injury. Participants' clinical status will be monitored until they no longer need ventilation and return home, or for up to 60 days while in the hospital. Individuals being treated for ARDS at the participating hospitals who decline to enroll in the study will be asked for permission to monitor their medical progress. These individuals will not take part in any study procedures, but their clinical information will be used for comparison purposes. Additionally, clinical information on other ARDS patients admitted to the hospital over the previous 2 years will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of all of the following criteria within a 24-hour period:

  1. Bilateral infiltrates consistent with edema on frontal chest radiograph, with a duration of no more than 7 days
  2. Requires positive pressure ventilation through an endotracheal tube
  3. PaO2/FiO2 less than 200 while receiving positive end-expiratory pressure (PEEP) at more than 8 cm H2O for at least 4 hours, with a duration of no more than 7 days
  4. No clinical evidence of left atrial hypertension

Exclusion Criteria:

* Weighs less than 35 kilograms
* Receives more than 5 days of mechanical ventilation during current hospitalization
* Attending physician declines to give consent for participant to enroll
* Patient or surrogate declines or is unable to give consent
* Participation in another interventional study for ARDS in the 30 days prior to study entry
* Intracranial hypertension
* Single lung transplant
* Burns over more than 30% of the surface area of the body
* Pregnant
* Sickle (Hgb SS) or sickle-thal (Hgb SC) hemoglobin
* Pre-existing illness with a life expectancy of 6 months or less
* Physicians and family are not committed to full support (Exception: An individual will not be excluded if he/she would receive all medical care except for attempts at resuscitation from cardiac arrest)
* Severe chronic lung disease
* Prior lung resection
* More than 72 hours has passed since inclusion criteria were met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of ventilator free days | Measured at 28 days
Changes in plasma concentration of IL-6 | Measured at 3 days

SECONDARY OUTCOMES:
Number of intensive care unit free days | Measured at 28 days
Mortality | Measured at 60 days
Number of hospital free days | Measured at 60 days
Changes in plasma IL1ra | Measured at 3 days
Changes in plasma IL-1 | Measured at 3 days
Changes in plasma IL-10 | Measured at 3 days
Changes in plasma surfactant protein D | Measured at 3 days
Changes in plasma von Willebrand factor | Measured at 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Roy G. Brower, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Ohio State University Medical Center, Columbus, Ohio
  - Wilford Hall Medical Center, San Antonio, Texas

REFERENCES:
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Krishnan JA, Brower RG. High-frequency ventilation for acute lung injury and ARDS. Chest. 2000 Sep;118(3):795-807. doi: 10.1378/chest.118.3.795. PMID 10988205
- [Background] Derdak S, Mehta S, Stewart TE, Smith T, Rogers M, Buchman TG, Carlin B, Lowson S, Granton J; Multicenter Oscillatory Ventilation For Acute Respiratory Distress Syndrome Trial (MOAT) Study Investigators. High-frequency oscillatory ventilation for acute respiratory distress syndrome in adults: a randomized, controlled trial. Am J Respir Crit Care Med. 2002 Sep 15;166(6):801-8. doi: 10.1164/rccm.2108052. PMID 12231488
- [Background] Randomized study of high-frequency oscillatory ventilation in infants with severe respiratory distress syndrome. HiFO Study Group. J Pediatr. 1993 Apr;122(4):609-19. doi: 10.1016/s0022-3476(05)83548-6. PMID 8463913